CLINICAL TRIAL: NCT01555242
Title: A Phase I, Open-Label, Multiple Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral Aneustat™ (OMN54) Administered on a Daily Oral Regimen in Patients With Advanced Cancer and Lymphomas
Brief Title: A Study of Aneustat (OMN54) in Patients With Advanced Cancer and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Omnitura Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMN54-101
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms
Keywords: Advanced Cancer; Lymphoma; Refractory
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aneustat (OMN54) (Experimental)
  Interventions: Drug: Aneustat (OMN54)

INTERVENTIONS:
Drug: Aneustat (OMN54) — 100 mg active/capsule; oral administration; 28 days/cycle (up to 6 cycles total) 1,000 mg QD 2,000 mg QD 1,500 mg BID 2,000 mg BID 2,500 mg BID

SUMMARY:
This is a phase I, open-label, multiple dose, dose escalation study to assess the safety, tolerability and pharmacokinetics of Aneustat™ (OMN54), a novel therapy, administered orally in patients with advanced cancer and lymphomas.

DETAILED DESCRIPTION:
Patients who complete a 28-day cycle, may be eligible to continue receiving Aneustat™ (OMN54) in 4-week increments for up to 6 cycles (inclusive of cycle 1) if further treatment is judged to be of possible benefit; if patient has not experienced unacceptable toxicity; and no study withdrawal criteria has been met.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of malignancy
* Male or female, 18 years or older
* Presence of advanced tumours, i.e., measurable or non-measurable disease (RECIST criteria, version 1.1)that have recurred or progressed following standard therapy
* Able to swallow the oral capsule form of the drug
* Failed at least one previous therapeutic regimen and either no longer are candidates for standard therapy, have no standard therapy available, or choose not to pursue standard therapy.
* Haematology within 7 days of Day 1 (initial dose):

  * Hemoglobin (Hb) > 9.0 g/dL
  * Platelets ≥ 100,000 cells/mm3 (or, ≥100 x 10/L)
  * Absolute neutrophil count (ANC) > 1.5 cells x109/L (or, > 1500 cells/mm3)
* Chemistry within 7 days of Day 1 (initial dose):

  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x ULN if no liver metastases, AST(SGOT)/ALT(SGPT) < 5 x ULN if liver metastases
  * Bilirubin < 1.5 x ULN unless Gilbert's Syndrome
  * Serum creatinine ≤ 1.25 ULN
* Coagulation within 7 days of Day 1 (initial dose):

  *INR ≤ 1.5
* ECOG Performance Status between 0 - 2 and estimated life expectancy of > 3 months.
* Having the initiative and means to be compliant with the protocol (as judged by the Principal Investigator) and is within a feasible geographical proximity of the study center to make the required study visits.
* Written informed consent obtained prior to any study screening procedures
* Females of childbearing potential (a female is considered of childbearing potential unless she is postmenopausal, i.e., no menses for at least 12 consecutive months, or is without a uterus) must have a negative urine pregnancy test (UPT) within 7 days of Day 1 (initial dose)
* Females of childbearing potential must agree to use an effective method of contraception (i.e., sexual abstinence, condoms, intrauterine device, diaphragm) from Screening period and throughout study participation.

Exclusion Criteria:

* Patient has uncontrolled or symptomatic brain metastases (If a patient has brain metastases and is on steroids, the steroid dose must be stable for at least 30 days prior to Day 1 dosing).
* Use of an investigational medication or device within 30 days of initiating study therapy (Day 1).
* Major surgery within 30 days prior to first dose (Day 1).
* Radiotherapy, chemotherapy, or immunotherapy within 28 days prior to Day 1 (not including palliative radiotherapy at focal sites).
* Pregnancy or lactation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NY Heart Association Class III or IV, see Appendix 3), unstable angina pectoris, unstable cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements.
* Screening (within approximately 28 days of registration) 12-lead electrocardiogram (ECG) that is abnormal and clinically significant
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* Use of warfarin, i.e., Coumadin®, Jantoven® within 7 days prior to Day 1 (initial dosing)
* Intolerance or aversion to porcine ingredients that are used for the OMN54 oral capsules in the investigational medicine, OMN54 (Aneustat™).
* Known hypersensitivity to any of the three botanical constituents of Aneustat™ (OMN54), or other similar plants; or to plants belonging to Labiatae or Lamiaceae families, soy, or Aneustat™ (OMN54) excipients
* Use of Sophora subprostrata root (SSR) or herba serissae within 14 days prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of two dosing regimens (once daily and twice daily)
  The maximum tolerated dose (MTD) is defined as the dose, based on data from 6 patients (or 5 patients if one patient has withdrawn due to non-Aneustat (OMN54) related reasons), below the non-tolerated dose (DL T).
Dose Limiting Toxicity (DLT) of two dosing regimens (once daily and twice daily)
  Assessment per Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Plasma blood concentrations of chemical markers
  These measurements are intended to characterize the pharmacokinetics of Aneustat (OMN54)

SECONDARY OUTCOMES:
Tumor Response
  Tumor response as per RECIST criteria version 1.1, and tumor markers in plasma, as applicable
Measurement of pathway biomarkers in plasma
  Plasma concentrations of cancer-related proteins to help characterize Aneustat (OMN54) activity

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Agency-Vancouver Centre, Vancouver, British Columbia, Canada